CLINICAL TRIAL: NCT06146166
Title: Prospective, Double-Blinded, Randomized Placebo Controlled Trial of an Oral Hair Supplement on Hair Density, Growth, and Microbiome
Brief Title: The Effects of an Oral Hair Supplement on Hair Density, Growth, and Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Vidya Herbs (Sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: i23-10-VIDYA_HAIR_SUPP
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hair Thinning
MeSH Terms: conditions — Alopecia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral herbal supplement (Experimental): Oral supplement containing an herbal blend
  Interventions: Dietary Supplement: Oral herbal supplement
- Oral Placebo Supplement (Placebo Comparator): Oral placebo supplement
  Interventions: Dietary Supplement: Oral placebo supplement

INTERVENTIONS:
Dietary Supplement: Oral herbal supplement — Oral supplement containing an oral blend taken once daily
  Arms: Oral herbal supplement
Dietary Supplement: Oral placebo supplement — Oral placebo supplement taken once daily
  Arms: Oral Placebo Supplement

SUMMARY:
The purpose of this study is to assess how an oral herbal supplement influences hair density, shine, growth, and microbiome.

DETAILED DESCRIPTION:
Hair thinning and hair loss are highly prevalent conditions affecting both men and women. Various factors can contribute to hair thinning and loss, including nutrition, medications, family history, and more. Overall, hair thinning and loss have a significant impact on quality of life and patients with these concerns have limited options. For example, minoxidil, finasteride, hair transplantations, and platelet rich plasma are effective options but each are paired with their own limitations. Thus, those with hair thinning or loss are increasingly turning to natural therapies shown to improve hair density and self-perceived hair thinning.

Nutrition is closely related to hair health, as evidenced by hair thinning and loss that occur with malnutrition or restrictive diets. Additionally, the hair follicle microbiome has been shown to modulate inflammation that exacerbates inflammatory scalp diseases, and ultimately hair thinning and hair loss.

Thus, an oral supplement that addresses nutrient deficiencies and targets the hair follicle microbiome could support hair health. In this study, we examine the effects of an herbal oral supplement on hair density, shine, and growth.

ELIGIBILITY:
Inclusion Criteria:

- Men and women between the ages of 25 years old and 65 years old with self-perceived hair thinning.

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners.
* Adults unable to consent.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Subjects with scarring forms of alopecia.
* Any history of procedures affecting hair growth, such as transplantation
* Any known allergy to any of the ingredients in the study product.
* Any laser treatments for hair growth in the past 3 months
* Use of any over-the-counter or pharmaceutical or dietary products known to affect hair growth
* Subjects unwilling to not alter hair color or style for the duration of the study.
* Subjects taking any hair growth oral supplementation within the past 3 months.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.
* Those who have been on an oral antibiotic within 1 month prior enrolling
* Those who are unwilling to discontinue oral probiotics-based supplementation or supplement ingredients found in the study's oral, product 1 month prior to enrollment

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Hair density | 24 weeks
  Change in hair density as measured by Trichogram based photographic analysis

SECONDARY OUTCOMES:
Hair density | 4 weeks
  Change in hair density as measured by Trichogram based photographic analysis
Hair diameter | 24 weeks
  Change in hair diameter and hair diameter
Hair diameter | 4 weeks
  Change in hair diameter and hair diameter
Shannon diversity of hair microbiome | 24 weeks
  Shift in Shannon diversity measure of the hair microbiome
Hair health measured by global photographs as subjective factors graded by the investigator | 4 weeks
  Change in hair growth, density, and shine measured by global photographs as subjective factors graded by the investigator
Hair health measured by global photographs as subjective factors graded by the investigator | 24 weeks
  Change in hair growth, density, and shine measured by global photographs as subjective factors graded by the investigator
Self-perception of hair | 4 weeks
  10-question survey based self grading of hair growth, density, and shine measured with subjective questionnaire. Answers range from Strongly Agree, Agree, Neutral, Disagree, or Strongly Disagree.
Self-perception of hair | 24 weeks
  10-question survey based self grading of hair growth, density, and shine measured with subjective questionnaire. Answers range from Strongly Agree, Agree, Neutral, Disagree, or Strongly Disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No